CLINICAL TRIAL: NCT00562939
Title: Immune Response to Toll-Like Receptor 9-Agonist Adjuvanted Pneumococcal Vaccination in HIV Infected Adults
Acronym: ITAP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Ole Søgaard, MD, Department of Infectious Diseases, Skejby
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2007-001588-31
Record Dates: First submitted 2007-11-23; First posted 2007-11-26 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: HIV Infections
Keywords: Antibody Formation; Antibody Affinity; Immunity; Pneumococcal Vaccines; Oligodeoxyribonucleotides
MeSH Terms: conditions — HIV Infections | interventions — Pneumococcal Vaccines; ProMune

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): 1 mg CpG 7909 + pneumococcal vaccines
  Interventions: Biological: Pneumococcal vaccines + CPG 7909
- B (Placebo Comparator): Pneumococcal vaccines
  Interventions: Biological: Pneumococcal vaccines

INTERVENTIONS:
Biological: Pneumococcal vaccines + CPG 7909 — Day 0: 1 ml Prevenar (double dose) + 1 mg CpG 7909, IM Day 90: 1 ml Prevenar (double dose) + 1 mg CpG 7909, IM Day 270: 0.5 ml Pneumo Novum + 1 mg CpG 7909, IM
  Other Names: Cpg 7909/Vaximmune(TM)
  Arms: A
Biological: Pneumococcal vaccines — Day 0: 1 ml Prevenar (double dose) + placebo, IM Day 90: 1 ml Prevenar (double dose) + placebo, IM Day 270: 0.5 ml Pneumo Novum + placebo, IM
  Arms: B

SUMMARY:
The purpose of this study is to determine whether TLR-9 adjuvanted pneumococcal is more immunogenic than pneumococcal vaccination alone in HIV-infected adults.

DETAILED DESCRIPTION:
Pneumococcal disease is a major source of morbidity and mortality in HIV-patients. HIV-patients are vaccine hyporesponders. A good immune response to pneumococcal vaccination enhances vaccine effectiveness, thereby preventing the morbidity and mortality caused by pneumococcal disease. Even when an optimized regimen containing both conjugated and polysaccharide pneumococcal vaccine is used, only 13% of the immunized HIV patients are high responders at week 96. Recent data indicate that TLR9-agonists have excellent vaccine adjuvant potential and are safe to use in immunocompetent as well as immunocompromised individuals. The aim of this study is to evaluate the qualitative and quantitive immune response to pneumococcal vaccination with or without TLR9-agonist in HIV-infected adults

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and authority statement provided according to local regulatory and ethical practice using a participant information sheet and informed consent form approved by the responsible Ethics Committee.
* HIV-seropositive individuals.

Exclusion Criteria:

* Pregnancy as determined by a positive urine beta-hCG (if female)
* Participant unwilling to use reliable contraception methods for the duration of the trial. Reliable methods of birth control include: pharmacologic contraceptives including oral, parenteral, and transcutaneous delivery; condoms with spermicide; diaphragm with spermicide; surgical sterilization; vaginal ring; intrauterine device; abstinence; and post-menopause (if female)
* Currently breast-feeding (if female)
* Latest CD4 count < 200 x106 cells/µL
* Viral load (HIV RNA) > 50 copies/mL if on HAART (defined as at least three antiretrovirals including either a protease inhibitor or a NNRTI, i.e. combivir 300/150 mg x2 + stocrin 600 mg x1 for a minimum of 6 months)
* Previous enrollment in this study
* Any medical, psychiatric, social, or occupational condition or other responsibility that, in the judgment of the Principal Investigator (PI), would interfere with the evaluation of study objectives (such as severe alcohol abuse, severe drug abuse, dementia)
* Unable to follow protocol regimen
* Pneumococcal vaccination 5 years or less prior to inclusion
* Planned participation in other vaccination trials during the time of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Numbers of vaccine high responders - defined as 2-fold increase and IgG levels ≥1 µg/mL to at least 5 of 7 pneumococcal serotypes (by quantitative IgG measurements) - in the CpG 7909 group vs. the control group | At day 270

SECONDARY OUTCOMES:
Functional activity of anticapsular antibodies measured by OPA | At day 90, 120, 270, 300
Safety/Tolerability | During the entire trial period
Nasopharyngeal pneumococcal colonization | At day 270
Predictors of antibody response, i.e. CD4+ cell count and sCD163 | At baseline
Numbers of vaccine high responders - defined as 2-fold increase and IgG levels ≥1 µg/mL to at least 5 of 7 pneumococcal serotypes (by quantitative IgG measurements) - in the CpG 7909 group vs. the control group | At day 90,120 and 300
Quantity and differentiation of IgG subtypes for HAART-experienced and HAART-naive individuals | Day 0, 90, 120
Cytokine response to various antigens by in vitro cell stimulation for HAART-experienced and HAART-naive individuals | At day 0, 90, 120

CONTACTS AND LOCATIONS:
Overall Officials: Ole Sogaard, MD, Principal Investigator — Department of Infectious Diseases, Aarhus University Hospital, Denmark; Lars Ostergaard, MD,PhD,DmSC, Study Director — Department of Infectious Diseases, Aarhus University Hospital, Denmark
Locations (1):
- Department of Infectious Diseases, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Offersen R, Melchjorsen J, Paludan SR, Ostergaard L, Tolstrup M, Sogaard OS. TLR9-adjuvanted pneumococcal conjugate vaccine induces antibody-independent memory responses in HIV-infected adults. Hum Vaccin Immunother. 2012 Aug;8(8):1042-7. doi: 10.4161/hv.20707. Epub 2012 Aug 1. PMID 22854665
- [Derived] Sogaard OS, Lohse N, Harboe ZB, Offersen R, Bukh AR, Davis HL, Schonheyder HC, Ostergaard L. Improving the immunogenicity of pneumococcal conjugate vaccine in HIV-infected adults with a toll-like receptor 9 agonist adjuvant: a randomized, controlled trial. Clin Infect Dis. 2010 Jul 1;51(1):42-50. doi: 10.1086/653112. PMID 20504165